CLINICAL TRIAL: NCT03089281
Title: Strategic Management to Optimize Response To Cardiac Resynchronization Therapy
Acronym: SMART CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C2067
Record Dates: First submitted 2017-03-19; First posted 2017-03-24 (Actual); Results first posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SmartDelay™ algorithm (Other): Subjects programmed with AV Delay and pacing chamber determined by SmartDelay
  Interventions: Device: CRT-D
- Fixed AV Delay with BiV pacing (Other): Subjects programmed with a Fixed AV Delay of 120ms with BiV pacing
  Interventions: Device: CRT-D

INTERVENTIONS:
Device: CRT-D — Commercially approved quadripolar Boston Scientific Cardiac Resynchronization Therapy Defibrillator (CRT-D) devices and future generations of BSC X4 CRT-D devices approved by the appropriate regulatory bodies will be included in the trial. All devices utilized in the study will include SmartDelay™ and must be capable of providing SmartDelay recommendations for both biventricular pacing (BiV) and Left Ventricular (LV) only pacing. All enrolled subjects with implanted BSC X4 CRT-D system and identified with an RV-LV delay of ≥70ms were 1:1 randomized. Randomization occurred in the electronic data capturing system.

SUMMARY:
The primary objective is to evaluate the benefit of the SmartDelay™ algorithm in patients with a prolonged RV-LV interval.

DETAILED DESCRIPTION:
The primary hypothesis of SMART CRT is that among cardiac resynchronization therapy defibrillator (CRT-D) patients with prolonged inrerventricular delay between the RV and LV leads, CRT with atrioventricular optimization (AVO) will result in greater reverse LV remodeling compared with CRT programmed at nominal settings (120 ms).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be indicated to receive a de novo quadripolar Boston Scientific Cardiac Resynchronization Therapy Defibrillator (CRT-D) in conjunction with an ACUITY X4 LV lead. This includes subjects who are indicated to receive an upgrade to a BSC X4 CRT-D from a previously implanted device.
* In order to achieve a homogenous population for the study, qualifying subjects are those with heart failure who meet BSC US indications for use defined as those subjects who receive stable optimal pharmacologic therapy (OPT) for heart failure and who meet any one of the following classifications:

  * Moderate to severe heart failure (NYHA Class III-IV) with EF ≤ 35% and QRS duration ≥ 120 ms
  * Left bundle branch block (LBBB) with QRS duration ≥ 130 ms, EF ≤ 30%, and mild (NYHA Class II) ischemic or nonischemic heart failure or asymptomatic (NYHA Class I) ischemic heart failure
* Subject is age 18 or above, or of legal age to give informed consent specific to each country and national laws
* Subject is willing and capable of providing informed consent
* Subject is willing and capable of complying with visits and procedures as defined by this protocol

Exclusion Criteria:

* Subjects with documented permanent complete AV block
* Subjects with permanent or chronic atrial fibrillation (AF) or in AF at the time of enrollment
* Subjects who have previously received cardiac resynchronization therapy with pacing in the left ventricle
* Subjects on the active heart transplant list or who has or is to receive ventricular assist device (VAD)
* Life expectancy shorter than 12 months due to any medical condition (e.g., cancer, uremia, liver failure, etc…)
* Subject with a known or suspected sensitivity to dexamethasone acetate (DXA)
* Subject is enrolled in any other concurrent clinical study, with the exception of local mandatory governmental registries and observational studies/registries, without the written approval from Boston Scientific
* Women of childbearing potential who are or plan to become pregnant during the course of the trial
* Subjects currently requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Gold, MD, Principal Investigator — Medical University of South Carolina
Locations (72):
- United States (41):
  - Affinity Hospital, LLC d/b/a Granview Medical Center, Birmingham, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - University of Arizona Sarver Heart Center, Tucson, Arizona
  - Cardiology Associates of NE Arkansas, Jonesboro, Arkansas
  - Glendale Adventist Medical Center, Glendale, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - Christiana Care Health Services, Newark, Delaware
  - Baptist Health Research Institute, Jacksonville, Florida
  - Watson Clinic Center for Research, Inc, Lakeland, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Heart Group at Deaconness Hospital, Newburgh, Indiana
  - University of Iowa Hospitals, Iowa City, Iowa
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Southcoast Health, Fall River, Massachusetts
  - Cardiovascular Institute of Michigan, Roseville, Michigan
  - Trinity Health Michigan d/b/a Michigan Heart, Ypsilanti, Michigan
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - The International Heart Institute on Montana Foundation, Missoula, Montana
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - The Ohio Health Research Institute- Grant Medical Center, Columbus, Ohio
  - Providence Heart Institute, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Pottstown Medical Specialist, Inc, Pottstown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - North Central Heart, Sioux Falls, South Dakota
  - Dallas VA Research Corporation, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Foundation for Advancing Veterans' Health Research, San Antonio, Texas
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
- Institut universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Canada
- France (7):
  - Centre hospitalier du pays d'Aix, Aix-en-Provence
  - CHU Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Hopital Saint Philibert, Lille
  - CHRU Hopital Pontchaillou, Rennes
  - Centre Hôpital Universitaire Rouen, Hôpital Charles Nicolle, Rouen
  - Centre Hôpital Universitaire Rangueil, Toulouse
- Germany (5):
  - Unfalkrankenhaus Marzahn, Berlin
  - University of Berlin, Charite Virchow Standort, Berlin
  - Uni Jena, Jena
  - Krankenhaus Landshut-Achdorf, Landshut
  - Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
- Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (2):
  - Ospedale S. Orsola - Malpighi, Bologna
  - Azienda Sanitaria Universtitaria Integrata di Trieste, Trieste
- Japan (4):
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Tokyo Medical University Hospital, Shinjuku-Ku, Tokyo
  - Shinshu University Hospital, Nagano
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Spain (3):
  - Hospital Infanta Cristina, Badajoz, Extremadura
  - Hospital 12 de Octubre Madrid, Madrid
  - Hospital Universitario La Fe, Valencia
- Cardiocentro Ticino, Lugano, Switzerland
- United Kingdom (6):
  - Royal Sussex County Hospital, Brighton
  - University Hospital of Wales, Cardiff
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospital, Nottingham
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Gold MR, Ellenbogen KA, Leclercq C, Lowy J, Rials SJ, Shoda M, Tomassoni G, Issa Z, Sarrazin JF, Jennings JM, Nair DG, Wold N, Yong P, Harbin MM, Stein KM, Auricchio A. Effects of Atrioventricular Optimization on Left Ventricular Reverse Remodeling With Cardiac Resynchronization Therapy: Results of the SMART-CRT Trial. Circ Arrhythm Electrophysiol. 2023 Jun;16(6):e011714. doi: 10.1161/CIRCEP.122.011714. Epub 2023 May 15. PMID 37183700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Commercially approved quadripolar Boston Scientific CRT-D devices and future generations of BSC X4 CRT-D devices approved by the appropriate regulatory bodies were included in the trial. All devices utilized in the study will include SmartDelay™ and must be capable of providing SmartDelay recommendations for both biventricular pacing (BiV) and Left Ventricular (LV) only pacing.
Pre-assignment Details: 699 subjects were enrolled. 259 were exited prior to randomization (88 not implanted, 7 no RV-LV measurement, 161 RV-LV < 70ms, 3 no viable pacing vector). Subjects with an RV-LV delay >= 70ms were randomized (n = 440). Randomized subjects received a Boston Scientific Cardiac Resynchronization Therapy Defibrillator (CRT-D) and were randomized 1:1 to have either an AV Delay and pacing chamber determined by SmartDelay or a Fixed AV Delay of 120ms with BiV pacing.
Groups:
- SmartDelay™ Algorithm: AV Delay and pacing chamber were determined by SmartDelay algorithm
- Fixed AV Delay With BiV Pacing: Fixed AV Delay of 120ms with BiV pacing was programmed
Period: Overall Study
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Started | 225 | 215
Completed | 197 | 198
Not Completed | 28 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing | Total
Number analyzed (Participants) | 225 | 215 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (10.6) | 67.6 (10.1) | 66.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 72 | 161
  Male | 136 | 143 | 279
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data not reported on 44 participants.
  Participants
    number analyzed (Participants) | 206 | 190 | 396
    Black or African Heritage | 30 | 22 | 52
    Caucasian | 160 | 155 | 315
    Hispanic or Latino | 12 | 9 | 21
    Asian | 3 | 3 | 6
    Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 134 | 123 | 257
  France | 18 | 19 | 37
  Canada | 15 | 16 | 31
  Germany | 14 | 16 | 30
  United Kingdom | 14 | 13 | 27
  Spain | 14 | 12 | 26
  Japan | 5 | 5 | 10
  Netherlands | 5 | 4 | 9
  Italy | 4 | 4 | 8
  Switzerland | 2 | 2 | 4
  Ireland | 0 | 1 | 1
New York Heart Association (NYHA) Classification [Count of Participants; unit: Participants] — The Stages of Heart Failure:
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 meters).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    Class I | 4 | 5 | 9
    Class II | 97 | 91 | 188
    Class III | 122 | 115 | 237
    Class IV | 2 | 4 | 6
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: % of blood ejected during LV contraction] — Population: LVEF data was unavailable for some participants due to missing measurement or unreadable echocardiogram data.
  % of blood ejected during LV contraction
    number analyzed (Participants) | 205 | 195 | 400
    (all) | 27.4 (9.9) | 28.0 (8.9) | 27.7 (9.4)
Left Ventricular End Systolic Volume (LVESV) [Mean (Standard Deviation); unit: milliliters] — Population: LVESV data was unavailable for some participants due to missing measurement or unreadable echocardiogram data.
  milliliters
    number analyzed (Participants) | 205 | 195 | 400
    (all) | 148 (64) | 140 (60) | 144 (62)
Conduction Disorder [Count of Participants; unit: Participants] — Population: Data not reported for one participant.
  Participants
    number analyzed (Participants) | 225 | 214 | 439
    Left Bundle Branch Block (LBBB) | 204 | 193 | 397
    Right Bundle Branch Block (RBBB) | 2 | 4 | 6
    Intraventricular Conduction Delay (IVCD) | 19 | 17 | 36
QRS width (ms) [Mean (Standard Deviation); unit: milliseconds] | 164 (20) | 160 (16) | 162 (18)

OUTCOME MEASURES:

1. Primary Outcome: CRT Response
Description: Comparing cardiac resynchronization therapy (CRT) response rates between AV Delay programming schemes defined by SmartDelay or a Fixed AV Delay of 120ms. A negative change in LVESV is considered an improvement; CRT response is defined by a change in Left Ventricular End Systolic Volume (LVESV) < -15% at 6 months compared to pre-implant baseline.
Time Frame: Pre-Implant baseline to 6 months
Population: A total of 130 randomized subjects did not contribute data to the primary endpoint analysis due to death or withdrawal prior to six months, missed six-month visit or incomplete/insufficient echocardiogram.
Measure: Count of Participants; unit: Participants
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 155 | 155
Participants | 116 | 105
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.17, Chi-squared

2. Secondary Outcome: Change in Left Ventricular End Systolic Volume (Absolute Change)
Description: Comparing absolute changes in Left Ventricular End Systolic Volume from Implant to 6 Months between AV Delay programming schemes defined by SmartDelay or a Fixed AV Delay of 120ms. Change is defined as 6-Month measurement - Implant measurement, in milliliters. A negative change in LVESV is considered an improvement.
Time Frame: Implant to 6 Months
Population: A total of 130 randomized subjects did not contribute data to the secondary endpoint analysis due to death or withdrawal prior to six months, missed six-month visit or incomplete/insufficient echocardiogram.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 155 | 155
milliliters | -51.5 (51.1) | -37.8 (42.3)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.011, t-test, 2 sided

3. Secondary Outcome: Change in Left Ventricular End Systolic Volume (Relative Change)
Description: Comparing relative changes in Left Ventricular End Systolic Volume from Implant to 6 Months between AV Delay programming schemes defined by SmartDelay or a Fixed AV Delay of 120ms. Change is defined as 100*(6-Month measurement - Implant measurement)/(Implant Measurement), in %. A negative change in LVESV is considered an improvement.
Time Frame: Implant to 6 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 155 | 155
% change | -33.2 (25.2) | -26.7 (27.4)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.029, t-test, 2 sided

4. Secondary Outcome: Change in Left Ventricular Ejection Fraction (Absolute Change)
Description: Comparing absolute changes in Left Ventricular Ejection Fraction from Implant to 6 Months between AV Delay programming schemes defined by SmartDelay or a Fixed AV Delay of 120ms. Change is defined as 6-Month measurement - Implant measurement, in % of blood ejected during LV contraction. A positive change in LVEF is considered an improvement.
Time Frame: Implant to 6 Months
Population: A total of 129 randomized subjects did not contribute data to the secondary endpoint analysis due to death or withdrawal prior to six months, missed six-month visit or incomplete/insufficient echocardiogram.
Measure: Mean (Standard Deviation); unit: % of blood ejected during LV contraction
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 155 | 156
% of blood ejected during LV contraction | 12.6 (11.5) | 10.2 (11.4)

5. Secondary Outcome: Change in Left Ventricular Ejection Fraction (Relative Change)
Description: Comparing relative changes in Left Ventricular Ejection Fraction from Implant to 6 Months between AV Delay programming schemes defined by SmartDelay or a Fixed AV Delay of 120ms. Change is defined as 100*(6-Month measurement - Implant measurement)/(Implant Measurement), in %. A positive change in LVEF is considered an improvement.
Time Frame: Implant to 6 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 155 | 156
% change | 57.5 (60) | 44.8 (54.2)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.050, t-test, 2 sided

6. Secondary Outcome: Clinical Composite Score (CCS)
Description: Th CCS combines four metrics: all-cause mortality, heart failure hospitalization (HFH), New York Heart Association (NYHA) Class, and quality of life as measured with the patient global assessment (GA) instrument.
  The CCS categorizes each subject into one of three groups: Improved, Unchanged or Worsened.
  * Improved: Subjects that survived without a HFH through the 6-month visit window and had either an improvement in NYHA class or responded to GA with "much better" or "very much better".
  * Unchanged: All patients that reached the end of 6-month visit window that were not categorized as either "Improved" or "Worsened".
  * Worsened: Subjects that died or had HFH within 6-month visit window or had either a worsening in NYHA class or responded to GA with "much worse" or "very much worse".
Time Frame: Implant to 6 Months
Population: Subjects that were followed through the end of the 6-month visit window and those that died and/or or had a heart failure hospitalization within the 6-month visit window contributed to this endpoint. A total of 34 subjects did not meet these conditions are were therefore excluded from endpoint analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 207 | 199
Participants
  Improved | 153 | 154
  Unchanged | 31 | 25
  Worsened | 23 | 20
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.49, Cochran-Armitage Trend Test

7. Secondary Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: The KCCQ is a disease-specific instrument for monitoring the health status and quality of life of subjects with congestive heart failure. It includes a total of 23 items that assess quality of life in the following domains: physical function, symptom frequency and severity, symptom stability, self-efficacy and knowledge, social function, and overall quality of life. These domains can be combined into a functional status summary score (derived from the physical function and symptom scales) and an overall summary score which combines the physical function, symptom, social function and quality of life domains.
  KCCQ scores have a minimum of 0 and a maximum of 100. Higher score indicates better quality of life.
Time Frame: Implant to 6 Months
Population: Subjects that completed the KCCQ at both the implant and 6 month visits contributed to this endpoint. A total of 51 subjects did not contribute data to the endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 194 | 195
score on a scale | 18.3 (21.0) | 20.2 (19.7)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.36, t-test, 2 sided

8. Other Pre Specified Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Social Limitation Score
Description: The KCCQ Social Limitation Domain quantifies the extent to which heart failure symptoms impair patients' ability to interact in a number of gender-neutral social activities.
  KCCQ scores have a minimum of 0 and a maximum of 100. Higher score indicates better quality of life.
Time Frame: Implant to 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 194 | 195
score on a scale | 17.1 (28.1) | 20.6 (25.1)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.21, t-test, 2 sided

9. Other Pre Specified Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Quality of Life Score
Description: KCCQ Quality of Life Domain is designed to reflect patients' assessment of their quality of life, given the current status of their heart failure.
  KCCQ scores have a minimum of 0 and a maximum of 100. Higher score indicates better quality of life.
Time Frame: Implant to 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 194 | 195
score on a scale | 25.0 (26.9) | 27.6 (26.3)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.34, t-test, 2 sided

10. Other Pre Specified Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Self-Efficacy Score
Description: KCCQ Self-efficacy Domain quantifies patients' perceptions of how to prevent heart failure exacerbations and manage complications when they arise. This scale is not included in the summary scores.
  KCCQ scores have a minimum of 0 and a maximum of 100. Higher score indicates better quality of life.
Time Frame: Implant to 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 194 | 195
score on a scale | 6.5 (21.8) | 4.9 (21.2)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.46, t-test, 2 sided

11. Other Pre Specified Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Symptom Frequency Score
Description: KCCQ Symptom Domain quantifies the frequency of clinical symptoms in heart failure, including fatigue, shortness of breath, paroxysmal nocturnal dyspnea and patients' edema/swelling.
  KCCQ scores have a minimum of 0 and a maximum of 100. Higher score indicates better quality of life.
Time Frame: Implant to 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 194 | 195
score on a scale | 15.6 (23.5) | 17.4 (23.2)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.45, t-test, 2 sided

12. Other Pre Specified Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Symptom Burden Score
Description: KCCQ Symptom Domain quantifies the burden of clinical symptoms in heart failure, including fatigue, shortness of breath, paroxysmal nocturnal dyspnea and patients' edema/swelling.
  KCCQ scores have a minimum of 0 and a maximum of 100. Higher score indicates better quality of life.
Time Frame: Implant to 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 194 | 195
score on a scale | 15.9 (23.5) | 15.6 (23.2)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.90, t-test, 2 sided

13. Other Pre Specified Outcome: Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) Physical Limitation Score
Description: KCCQ Physical Function Domain measures the limitations patients experience, due to their heart failure symptoms, in performing routine activities. Activities are common, gender-neutral, and generalizable across cultures, while also capturing a range of exertional requirements.
  KCCQ scores have a minimum of 0 and a maximum of 100. Higher score indicates better quality of life.
Time Frame: Implant to 6 Months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
Number analyzed (Participants) | 194 | 195
score on a scale | 14.6 (23.0) | 15.9 (23.2)
Statistical Analysis 1: Comparison: SmartDelay™ Algorithm vs Fixed AV Delay With BiV Pacing; Test type: Superiority; p = 0.59, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire duration of subject participation in the study. Subjects were followed for median of 6.5 months.
Arm/Group | SmartDelay™ Algorithm | Fixed AV Delay With BiV Pacing
All-Cause Mortality (participants affected / at risk) | 7/225 | 0/215
Serious Adverse Events (participants affected / at risk) | 49/225 | 46/215
Other Adverse Events (participants affected / at risk) | 20/225 | 22/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartDelay™ Algorithm (N=225) | Fixed AV Delay With BiV Pacing (N=215)
Infection > 30 Days Post-Implant (Pulse Generator-related) (Product Issues) | 2 | 0
Unable to Capture (Right Atrial Lead-related) (Product Issues) | 0 (0) | 1 (1)
Dislodgment (Right Atrial Lead-Related) (Product Issues) | 0 (0) | 1 (1)
Dislodgment (Right Ventricular Lead-Related) (Product Issues) | 1 (1) | 0 (0)
Dislodgment (Left Ventricular Lead-Related) (Product Issues) | 5 (5) | 4 (4)
Post-Surgical Wound Discomfort/Bruising/Swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-Surgical Infection (<=30 Days Post-Implant) (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Adverse Reaction - General (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hematoma - Pocket (<=30 Days Post-Implant) (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Thromboembolic Events (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Venous Occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart Failure (Cardiac disorders) | 14 (17) | 16 (24)
Ventricular Fibrillation (Cardiac disorders) | 3 (3) | 2 (2)
Ventricular Tachycardia/Monomorphic VT (Cardiac disorders) | 1 (1) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 2 (3) | 1 (1)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension/Orthostatic Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disease (Cardiac disorders) | 0 (0) | 2 (2)
Mitral Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Valvular Damage/Valvular Insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Dizziness (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain - Ischemic (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnea (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (CVA) (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Cardiac disorders) | 1 (1) | 2 (2)
Intracardiac Thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Septal Defect (Cardiac disorders) | 0 (0) | 1 (1)
Adverse Reaction - General (General disorders) | 1 (1) | 0 (0)
Adverse reaction - Allergic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Adverse reaction - Medication (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Systemic Infection (Infections and infestations) | 1 (1) | 3 (3)
Fever/Virus (General disorders) | 0 (0) | 1 (1)
Physical Trauma (General disorders) | 3 (3) | 3 (5)
Abnormal Laboratory Values (General disorders) | 1 (1) | 1 (2)
Neurological (General disorders) | 2 (2) | 2 (2)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 6 (6) | 4 (4)
Renal (Renal and urinary disorders) | 4 (6) | 2 (3)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Psychological (Psychiatric disorders) | 0 (0) | 1
Integumentary (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Endocrine (Endocrine disorders) | 1 (1) | 0 (0)
Immune (Immune system disorders) | 0 (0) | 1 (1)
Cancer (General disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SmartDelay™ Algorithm (N=225) | Fixed AV Delay With BiV Pacing (N=215)
Oversensing (Pulse Generator-related) (Product Issues) | 0 (0) | 1 (1)
Inappropriate Tachy Therapy (Pulse Generator-Related) (Product Issues) | 2 (2) | 1 (1)
Fatigue (Pulse Generator-Related) (Product Issues) | 1 (1) | 0 (0)
Dislodgment (Right Atrial Lead-Related) (Product Issues) | 1 (1) | 1 (1)
Dislodgment (Right Ventricular Lead-Related) (Product Issues) | 0 (0) | 1 (1)
Extracardiac Stimulation (Right Ventricular Lead-Related) (Product Issues) | 1 (1) | 0 (0)
Inappropriate Tachy Therapy (Right Ventricular Lead-Related) (Product Issues) | 0 (0) | 1 (1)
Unable to Capture (Left Ventricular Lead-Related) (Product Issues) | 2 (2) | 2 (2)
Extracardiac Stimulation (Left Ventricular Lead-Related) (Product Issues) | 4 (4) | 7 (7)
Perforation at Implant (Left Ventricular Lead-Related) (Product Issues) | 1 (1) | 0 (0)
Dislodgment (Left Ventricular Lead-Related) (Product Issues) | 2 (2) | 3 (3)
Hematoma - Pocket (<=30 days post-implant) (Surgical and medical procedures) | 1 (1) | 1 (1)
Pneumothorax (Surgical and medical procedures) | 1 (1) | 0 (0)
Lower Extremity Edema (Surgical and medical procedures) | 0 (0) | 1 (1)
Heart Failure (Cardiac disorders) | 3 (7) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Tachycardia / Other Supraventricular Tachycardia (SVT) (Cardiac disorders) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Fatigue / Weakness (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT03089281/Prot_SAP_000.pdf